CLINICAL TRIAL: NCT03201510
Title: HPTN 075: Feasibility of HIV Prevention Cohort Studies Among Men Who Have Sex With Men in Sub-Saharan Africa
Brief Title: Feasibility of HIV Prevention Cohort Studies Among Men Who Have Sex With Men in Sub-Saharan Africa
Status: Completed | Type: Observational
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: HPTN 075; UM1AI068619 (NIH)
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2022-08

CONDITIONS: HIV
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will be stored from each study visit
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational: Observational study
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — HPTN 075 is an observational study in sub-Saharan MSM

SUMMARY:
This study aims to determine the feasibility of recruiting and retaining men who have sex with men (MSM) in a multi-country prospective cohort study in preparation for human immunodeficiency virus (HIV) prevention studies in sub-Saharan Africa (SSA).

DETAILED DESCRIPTION:
HPTN 075 is an observational cohort study. Participants will be accrued over six months at four sites in SSA using convenience sampling strategies, with no replacement for participants lost to follow-up. Each participant will be followed for 12 months, during which five study visits involving structured HIV behavioral assessments, medical examinations, and collection of biological samples will be conducted (including enrollment and quarterly follow-up visits). Participants who do not complete 12 months of follow-up will be contacted to explore reasons for no longer participating.

ELIGIBILITY:
Inclusion Criteria:

* Biologically male at birth, according to self-report;
* 18-44 years old (inclusive);
* Willing and able to provide informed consent;
* Willing to undergo HIV testing throughout the study and to receive those test results;
* Reporting at least one act of anal intercourse in the previous 3 months (12 weeks) with a person reported by the participant to be biologically male;
* Able to provide complete locator identification for themselves and at least two other personal contacts;
* Willing to participate in all scheduled study assessments, including specimen collection, laboratory assessments, and sample storage;
* Committing to not participate in any HIV intervention or vaccine study while participating in HPTN 075;
* Planning to remain in the study area for at least one year;
* For HIV-uninfected men: All HIV test results at the Screening visit must be non-reactive/negative;
* For HIV-infected men (up to 20 per site): All HIV test results at the Screening visit must be reactive/positive.

Men who are already on PrEP will not be excluded. Additionally, self- or other-identified transgender women and male sex workers will not be excluded. There will, however, be no specific effort to recruit these groups.

Exclusion Criteria:

* Unwilling to adhere to study procedures;
* Past or current participation in a biomedical and/or behavioral HIV/STI intervention or cohort study, including HIV vaccine studies; however, participation in local/area PrEP demonstration projects does not preclude participation in HPTN 075;
* HIV-infected men who report that they are already on ART or in HIV care;
* Any other reason or condition that in the opinion of the Investigator of Record (IOR) would interfere with participation, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* Men who have discordant HIV test results at Screening (i.e., at least one reactive or positive result and at least one non-reactive or negative result). These men will receive HIV counseling and will be referred for further diagnostic tests and care.

Ages: 18 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men, regardless of HIV infection status, aged 18-44 years living in SSA who report anal sex with a man in the past 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2017-08-12 (Actual)

PRIMARY OUTCOMES:
Recruitment of approximately 400 participants | July 2015-July 2016
  all 4 sites must collectively recruit 400 participants
Retention of approximately 400 participants | July 2015-July 2016
  at least 90% of participants must be retained

SECONDARY OUTCOMES:
HIV incidence | July 2015-July 2017
  Measured by HIV RNA from plasma samples

CONTACTS AND LOCATIONS:
Overall Officials: Theodorus Sandfort, PhD, Study Chair — Columbia University
Locations (4):
- Kisumu, Kisumu, Kenya
- Johns Hopkins Project, Blantyre, Chichiri, Malawi
- South Africa (2):
  - Groote Schuur, Observatory, Cape Town
  - PHRU, Soweto, Gauteng

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT03201510/Prot_ICF_000.pdf